CLINICAL TRIAL: NCT02405208
Title: A Multi-center Outcomes Clinical Study of the PyroTITAN™ HRA Shoulder Implant in Humeral Head Resurfacing
Acronym: CHRA
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-HRA-002
Record Dates: First submitted 2014-11-04; First posted 2015-04-01 (Estimated); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2024-11

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary cohort: Primary cohort will receive the PyroTITAN HRA device
  Interventions: Device: PyroTITAN HRA

INTERVENTIONS:
Device: PyroTITAN HRA — Humeral resurfacing using the PyroTITAN HRA device

SUMMARY:
This study is designed as a multi-center, nonrandomized, uncontrolled, unblinded, prospective clinical outcomes investigation to evaluate the short, mid and long term performance of the PyroTITAN™ HRA Shoulder prosthesis humeral replacement.

DETAILED DESCRIPTION:
This study is designed as a multi-center, nonrandomized, uncontrolled, unblinded, prospective clinical outcomes investigation to evaluate the short, mid and long term performance of the PyroTITAN™ HRA Shoulder prosthesis humeral replacement. The PyroTITAN™ HRA Shoulder prosthesis device configuration will include humeral resurfacing CAP without cement. Patients will be selected for recruitment into the study based upon the normally accepted criteria for primary shoulder resurfacing arthroplasty.

The investigation will be conducted by up to 10 International surgeons experienced in HRA. 387 subjects with PyroTITAN™ HRA Shoulder prosthesis arthroplasties will be implanted and followed for 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients selected for inclusion will present for primary shoulder surface replacement or arthroplasty with any of the following diagnoses:

   * Osteoarthritis
   * Rheumatoid / Inflammatory Arthritis
   * Post-traumatic arthritis.
   * Focal and large (Hill-Sachs) osteochondral defects.
2. Subject is able to or capable of providing consent to participate in the clinical investigation.
3. Subject agrees to comply with this protocol, including participating in required follow-up visits at the investigations site and completing study questionnaires.
4. Subject is at least 21 years of age and skeletally mature at the time of surgery.

Exclusion Criteria:

1. Have destruction of the proximal humerus to preclude rigid fixation of the humeral component.
2. Insufficient bone quality as determined by intra-operative evaluation.
3. Have arthritis with defective rotator cuff.
4. Have had a failed rotator cuff surgery.
5. Have loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
6. Have evidence of active infection.
7. Present with a condition of neuromuscular compromise of the shoulder (e.g., neuropathic joints or brachioplexis injury with a flail shoulder joint).
8. Are unwilling or unable to comply with a rehabilitation program or would fail to return for the postoperative follow-up visits prescribed by the protocol.
9. Are skeletally immature.
10. Have a known allergic reaction to pyrocarbon.
11. Have other conditions such as central nervous system disturbances, alcohol or drug addiction, etc. that may make effective evaluation of the joint replacement difficult or impossible.
12. Are currently participating in another clinical study.
13. Have known, active metastatic or neoplastic disease.
14. Are taking > 10mg/day corticosteroids (e.g. prednisone) excluding inhalers, within 3 months prior to surgery.
15. Are under 21 years of age or over 75.

    .
16. Require glenoid replacement (Glenoid Classification).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who require humeral head resurfacing arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lankiewicz, Study Director — Smith & Nephew, Inc.
Locations (5):
- Australia (2):
  - Brisbane Hand & Upper Limb Clinic, Brisbane, Queensland
  - Barwon Health, Geelong, Victoria
- Institut Nices, Nice, France
- Danderyd Hospital, Stockholm, Sweden
- Wrightington Hospital, Wigan, Wrightington, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 156 participants were enrolled to the study at five (5) sites.
Pre-assignment Details: The Full Analysis Set (FAS) population includes 10 participants that received the TITAN device and 146 participants that received the PyroTITAN device. The TITAN device was renamed PyroTITAN by the previous sponsor (i.e., the same device). All participants were enrolled the same based on the eligibility criteria, so all participants are combined under the same primary cohort.
Groups:
- Primary Cohort: Primary cohort will receive the PyroTITAN HRA device*
  PyroTITAN HRA: Humeral resurfacing using the PyroTITAN HRA or TITAN device.
Period: Overall Study
Arm/Group | Primary Cohort
Started | 156
Completed | 73
Not Completed | 83

BASELINE CHARACTERISTICS:
Population: Full Analysis Set Population (FAS), following Intent-to-Treat principle included all participants enrolled into the study with data collected. This population includes 10 participants that received the TITAN device and 146 participants that received the PyroTITAN device. The TITAN device was renamed PyroTITAN by the previous sponsor (i.e., the same device). All participants were enrolled the same based on the eligibility criteria, so all participants are combined under the same primary cohort.
Groups:
- Primary Cohort: Primary cohort will receive the PyroTITAN HRA device
  PyroTITAN HRA: Humeral resurfacing using the PyroTITAN HRA or TITAN device
Arm/Group | Primary Cohort
Number analyzed (Participants) | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 102
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number of participants analyzed indicated participants with data collected for the baseline measure specified.
  kg/m^2
    number analyzed (Participants) | 153
    (all) | 29.00 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Device Survival
Description: Clinical success was determined by the percentage of shoulders with device survival. Survival of the device was measured by the Kaplan-Meier survival estimate with survival defined as all the following:
  * Device remained implanted
  * Absence of device-related complications requiring surgical replacement, removal, or augmentation of components
  * Freedom from chronic dislocation
Time Frame: up to 117 months
Population: Full Analysis Set Population (FAS) followed the Intent-to-Treat principle that included all participants enrolled with data collected for the outcome and time frame specified. Ten (10) participants received the TITAN device instead of the PyroTITAN device. These 10 participants were included in the FAS population as they were enrolled similarly to all other participants.
Measure: Number (95% Confidence Interval); unit: percentage of shoulders
Units Other Than Participants: shoulders
Arm/Group | Primary cohort
Number analyzed (Participants) | 72
Number analyzed (shoulders) | 72
percentage of shoulders | 85.97 [79.76 to 92.19]

2. Secondary Outcome: Radiographic Success
Description: Radiographic success determined by:
  * No evidence of device failure, specifically progressive migration or implant loosening
  * Anatomic alignment is a criterion that may be included in the definition of success in some investigations
Time Frame: 2 years, 3 years, 4 years, 5 years, 8 years and 10 years
Population: Radiographic outcome data were not collected during the study period by the original sponsor, despite being specified in the protocol. As a result, this outcome measure could not be analyzed or reported. This limitation does not affect the reporting of other pre-specified primary and secondary outcomes, which have been summarized and submitted as per protocol.
Arm/Group | Primary cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: ASES Score
Description: The ASES Shoulder Score is a functional outcome tool that has been validated for various shoulder conditions. ASES score ranges from 0 to 100, with a score of 0 indicating a worse shoulder condition and 100 indicating the best shoulder condition.
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary cohort
Number analyzed (Participants) | 153
score on a scale
  Baseline | 36.2 (16.1)
  3 months: number analyzed (Participants) | 151
  3 months | 66.0 (18.3)
  6 months: number analyzed (Participants) | 147
  6 months | 78.3 (18.4)
  1 year: number analyzed (Participants) | 142
  1 year | 82.5 (17.8)
  2 years: number analyzed (Participants) | 133
  2 years | 86.0 (17.6)
  3 years: number analyzed (Participants) | 108
  3 years | 85.7 (17.4)
  4 years: number analyzed (Participants) | 96
  4 years | 87.4 (15.8)
  5 years: number analyzed (Participants) | 119
  5 years | 86.5 (17.2)
  8 years: number analyzed (Participants) | 54
  8 years | 87.5 (20.2)
  10 years: number analyzed (Participants) | 69
  10 years | 89.3 (12.6)

4. Secondary Outcome: Visual Analog Scale (VAS) Pain Score
Description: The Visual Analog Scale (VAS) Pain Score ranges from 0 to 100, with 0 representing no pain (i.e., the best outcome) and 100 representing the worst possible pain (i.e., the worst outcome).
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary cohort
Number analyzed (Participants) | 154
score on a scale
  Baseline | 64.1 (20.3)
  3 months: number analyzed (Participants) | 151
  3 months | 24.2 (21.1)
  6 months: number analyzed (Participants) | 147
  6 months | 18.1 (20.2)
  1 year: number analyzed (Participants) | 143
  1 year | 15.5 (19.5)
  2 years: number analyzed (Participants) | 133
  2 years | 13.2 (19.4)
  3 years: number analyzed (Participants) | 110
  3 years | 15.5 (21.2)
  4 years: number analyzed (Participants) | 100
  4 years | 12.1 (18.1)
  5 years: number analyzed (Participants) | 124
  5 years | 13.4 (19.6)
  8 years: number analyzed (Participants) | 59
  8 years | 12.7 (21.9)
  10 years: number analyzed (Participants) | 72
  10 years | 9.2 (12.0)

5. Secondary Outcome: Visual Analog Scale (VAS) Satisfaction Score
Description: Patient satisfaction determined by the Visual Analog Scale (VAS) Satisfaction score. VAS Satisfaction scores range from 0 to 100, with 0 representing the lowest level of satisfaction (i.e., the worst possible outcome) and 100 representing the highest level of satisfaction (i.e., the best possible outcome).
Time Frame: 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary cohort
Number analyzed (Participants) | 151
score on a scale
  3 months | 75.8 (25.1)
  6 months: number analyzed (Participants) | 146
  6 months | 81.1 (23.3)
  1 year: number analyzed (Participants) | 143
  1 year | 84.0 (21.8)
  2 years: number analyzed (Participants) | 133
  2 years | 85.6 (21.8)
  3 years: number analyzed (Participants) | 110
  3 years | 85.6 (19.6)
  4 years: number analyzed (Participants) | 100
  4 years | 86.3 (18.5)
  5 years: number analyzed (Participants) | 124
  5 years | 86.1 (21.3)
  8 years: number analyzed (Participants) | 59
  8 years | 86.2 (24.2)
  10 years: number analyzed (Participants) | 72
  10 years | 88.6 (18.0)

6. Secondary Outcome: The Western Ontario of the Shoulder Index (WOOS) Score
Description: The WOOS Score is a quality of life questionnaire that has been validated for various shoulder conditions. WOOS total score ranges from 0 to 100, with 0 representing the best shoulder condition and 100 representing the worst shoulder condition.
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary cohort
Number analyzed (Participants) | 154
score on a scale
  Baseline | 65.1 (15.0)
  3 months: number analyzed (Participants) | 151
  3 months | 34.3 (19.9)
  6 months: number analyzed (Participants) | 146
  6 months | 22.2 (19.2)
  1 year: number analyzed (Participants) | 142
  1 year | 18.6 (19.5)
  2 years: number analyzed (Participants) | 134
  2 years | 15.3 (19.3)
  3 years: number analyzed (Participants) | 110
  3 years | 15.2 (17.0)
  4 years: number analyzed (Participants) | 100
  4 years | 14.2 (16.8)
  5 years: number analyzed (Participants) | 124
  5 years | 13.8 (15.6)
  8 years: number analyzed (Participants) | 58
  8 years | 12.6 (19.9)
  10 years: number analyzed (Participants) | 72
  10 years | 11.8 (13.9)

7. Secondary Outcome: Constant-Murley (CM) Score
Description: The Constant-Murley (CM) Score is a commonly used score of shoulder function. CM scores range from 0 to 100, with a score of 0 indicating a worse shoulder function (i.e., worst outcome) and 100 indicating the best shoulder function (i.e., best outcome).
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
Population: Full Analysis Set Population (FAS) followed the Intent-to-Treat principle that included all participants enrolled with data collected for the outcome and time frame specified. Ten (10) participants received the TITAN device instead of the PyroTITAN device. These 10 participants were included in the FAS population as they were enrolled similarly to all other participants. Data for 19 participants at 1 site excluded from analysis because data collection occurred using an incorrect CM format.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary cohort
Number analyzed (Participants) | 132
score on a scale
  Baseline | 39.4 (17.6)
  3 months: number analyzed (Participants) | 131
  3 months | 57.3 (18.8)
  6 months: number analyzed (Participants) | 127
  6 months | 72.5 (17.7)
  1 year: number analyzed (Participants) | 126
  1 year | 78.8 (16.0)
  2 years: number analyzed (Participants) | 116
  2 years | 82.5 (13.4)
  3 years: number analyzed (Participants) | 107
  3 years | 81.5 (14.1)
  4 years: number analyzed (Participants) | 91
  4 years | 82.1 (12.1)
  5 years: number analyzed (Participants) | 102
  5 years | 82.8 (12.3)
  8 years: number analyzed (Participants) | 54
  8 years | 83.4 (12.4)
  10 years: number analyzed (Participants) | 50
  10 years | 80.9 (11.6)

8. Secondary Outcome: EQ-5D-3L Quality of Life Score
Description: The EuroQol 5-Dimension 3-Level (EQ-5D-3L) Quality of Life Score ranges on a scale of 0 to 1, with 0 indicating a worse health condition (i.e., worst outcome) and 1 indicating the best health condition (i.e., best outcome).
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary cohort
Number analyzed (Participants) | 154
score on a scale
  Baseline | 0.759 (0.087)
  3 months: number analyzed (Participants) | 151
  3 months | 0.824 (0.097)
  6 months: number analyzed (Participants) | 147
  6 months | 0.860 (0.098)
  1 year: number analyzed (Participants) | 143
  1 year | 0.886 (0.098)
  2 years: number analyzed (Participants) | 134
  2 years | 0.870 (0.101)
  3 years: number analyzed (Participants) | 110
  3 years | 0.883 (0.100)
  4 years: number analyzed (Participants) | 100
  4 years | 0.887 (0.105)
  5 years: number analyzed (Participants) | 125
  5 years | 0.886 (0.114)
  8 years: number analyzed (Participants) | 59
  8 years | 0.888 (0.132)
  10 years: number analyzed (Participants) | 72
  10 years | 0.877 (0.121)

9. Secondary Outcome: EQ-5D-3L VAS Score
Description: The EuroQol 5-Dimension 3-Level (EQ-5D-3L) Visual Analog Scale (VAS) Score ranges on a scale of 0 to 100, with 0 indicating a worse health condition (i.e., worst outcome) and 100 indicating the best health condition (i.e., best outcome).
Time Frame: Baseline, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years, 8 years, and 10 years
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary cohort
Number analyzed (Participants) | 154
score on a scale
  Baseline | 61.9 (23.7)
  3 months: number analyzed (Participants) | 150
  3 months | 69.0 (19.0)
  6 months: number analyzed (Participants) | 147
  6 months | 71.3 (21.7)
  1 year: number analyzed (Participants) | 141
  1 year | 75.7 (17.6)
  2 years: number analyzed (Participants) | 134
  2 years | 75.2 (16.4)
  3 years: number analyzed (Participants) | 109
  3 years | 70.6 (22.0)
  4 years: number analyzed (Participants) | 99
  4 years | 71.9 (19.4)
  5 years: number analyzed (Participants) | 124
  5 years | 72.7 (22.3)
  8 years: number analyzed (Participants) | 58
  8 years | 76.8 (17.9)
  10 years: number analyzed (Participants) | 71
  10 years | 73.2 (18.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected upon implantation of the study device to the end of study, up to 10 years.
Description: Ascension Orthopedics Inc. conducted monitoring & reporting responsibilities from study start to December 2020. Upon acquisition, Smith+Nephew's Adverse Event Monitoring Board (AEMB) reviewed & classified all adverse events from January 2021 to the end of study, following ISO 14155 guidelines. It is unknown how the previous sponsor classified adverse events. 10 participants that received the TITAN device are combined with PyroTITAN due to renaming of the device as explained in Participant Flow.
Arm/Group | Primary Cohort
All-Cause Mortality (participants affected / at risk) | 7/156
Serious Adverse Events (participants affected / at risk) | 51/156
Other Adverse Events (participants affected / at risk) | 36/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort (N=156)
ABDOMINAL HERNIA (Surgical and medical procedures) | 1
AGGRAVATION OF HERNIATED DISC (General disorders) | 1
ANGINA ON EXERTION (Cardiac disorders) | 1
ARRHYTHMIA (Cardiac disorders) | 2
ARTHRITIS IN LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
ARTHRITIS IN RT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
BENIGN TUMOUR IN RIGHT KNEE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
BILATERAL ROTATOR CUFF DEGENERATION (Musculoskeletal and connective tissue disorders) | 1
BROKEN LEFT WRIST (Musculoskeletal and connective tissue disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC ARRHYTHMIA (Cardiac disorders) | 1
CHEST PAIN ON EXERTION (Cardiac disorders) | 1
CRACK IN PROSTHESIS (Product Issues) | 1
CUT ON LEFT INDEX FINGER USING DROP SAW (General disorders) | 1
DEVICE BREAKAGE (Product Issues) | 1
DIVERTICULITIS (Gastrointestinal disorders) | 1
FRACTURE IN HEAD OF IMPLANT (Product Issues) | 1
FRACTURE OF PYROTITAN IMPLANT (Product Issues) | 1
FRACTURED IMPLANT/PYROTITAN (Product Issues) | 1
GALL STONES (Renal and urinary disorders) | 1
IMPLANT BREAKAGE (Product Issues) | 2
IMPLANT BREAKAGE RIGHT SHOULDER (Product Issues) | 1
IMPLANT FRACTURE DUE TO A FALL (Product Issues) | 1
INCREASING LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1
INFLUENZA A (Infections and infestations) | 1
INFLUENZA TYPE A (Infections and infestations) | 1
KIDNEY STONES (Renal and urinary disorders) | 2
LEFT ELBOW PAIN (Musculoskeletal and connective tissue disorders) | 1
MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MELANOMA (CLARKS LEVEL 4) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MELANOMA (LEFT BIG TOE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MULTIPLE SCLEROSIS (Nervous system disorders) | 1
NECTROTISING INFLAMMATION OF RIGHT LUNG (Infections and infestations) | 1
NERVE PAIN IN LOWER BACK EXACERBATED (Musculoskeletal and connective tissue disorders) | 1
ONGOING LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1
PERSISTENT PAIN IN RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
PROSTATE INFECTION (Renal and urinary disorders) | 1
RADIAL NERVE PALSY (Nervous system disorders) | 1
REACTION TO IV DYE (General disorders) | 1
REFLUX (Gastrointestinal disorders) | 1
REVERSE TOTAL PROSTESIS LEFT SHOULDER (Product Issues) | 1
RIGHT ELBOW PAIN (Musculoskeletal and connective tissue disorders) | 1
RIGHT HAND CARPAL TUNNEL SYNDROME (Musculoskeletal and connective tissue disorders) | 1
RIGHT HIP BURSITIS (Musculoskeletal and connective tissue disorders) | 1
RIGHT KNEE PAIN / MENISCUS TEAR (Cardiac disorders) | 1
RIGHT ROTATOR CUFF INJURY (Musculoskeletal and connective tissue disorders) | 1
RIGHT ROTATOR CUFF TENDONITIS (Musculoskeletal and connective tissue disorders) | 1
RIGHT SHOULDER TENDINOPATHY (Musculoskeletal and connective tissue disorders) | 2
RUPTURED SPINAL DISCS (Musculoskeletal and connective tissue disorders) | 2
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1
STAGE 3 CHRONIC KIDNEY DISEASE. (Renal and urinary disorders) | 1
STAPH INFECTION IN RIGHT FOREARM (Infections and infestations) | 1
STONE IN GALL BLADDER (Renal and urinary disorders) | 1
STROKE (Vascular disorders) | 1
STROKE (Nervous system disorders) | 1
STROKE ATTACK (Nervous system disorders) | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
TIA (Vascular disorders) | 1
TORN RETINA IN RIGHT EYE (Eye disorders) | 1
TRAUMA TO THE LEFT KNEE. (Musculoskeletal and connective tissue disorders) | 1
WORSENING (R) SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1
WORSENING ARTHRITIS IN RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
WORSENING ARTHRITIS PAIN LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
WORSENING KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1
WORSENING KNEE PAIN (CATCHING) (Musculoskeletal and connective tissue disorders) | 1
WORSENING OA IN LEFT AND RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
WORSENING OA IN LEFT AND RIGHT KNEE due to BILATERAL TOTAL KNEE REPLACEMENT (Musculoskeletal and connective tissue disorders) | 1
WORSENING OA IN LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1
WORSENING OA RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF BILATERAL KNEE OA (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF LEFT KNEE OA. (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF LEFT KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF LEFT SHOULDER OA (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF OA IN LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 2
WORSENING OF OA IN RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF OA IN RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 2
WORSENING OF OA IN RIGHT THUMB (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF PRE-EXISTING BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF PRE-EXISTING HERNIA (General disorders) | 1
WORSENING OF RIGHT KNEE PAIN/ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF RIGHT SHOULDER OA. (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1
WORSENING OSTEOARTHRITIS IN LEFT KNEE (Musculoskeletal and connective tissue disorders) | 1
WORSENING PAIN IN RIGHT KNEE (Musculoskeletal and connective tissue disorders) | 1
WORSENING R) HIP OA (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Cohort (N=156)
AXILLARY NERVE DAMAGE RIGHT SHOULDER (Nervous system disorders) | 1
CUFF TENDINITIS IN RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
ONGOING PAIN IN LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 2
INCREASED PAIN IN OPERATIVE SHOULDER (Musculoskeletal and connective tissue disorders) | 1
LEFT SHOULDER NERVE IMPINGEMEN (Musculoskeletal and connective tissue disorders) | 1
PERSISTENT RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1
LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1
SEVERE INCREASE IN LEFT SHOULDER PAIN. (Musculoskeletal and connective tissue disorders) | 1
LEFT ROTATOR CUFF TENDONITIS (Musculoskeletal and connective tissue disorders) | 1
MARGINAL OSTEOPHYTE R GLENOID (Musculoskeletal and connective tissue disorders) | 1
CYSTIC CHANGES IN GLENOID NOTED ON MRI (Musculoskeletal and connective tissue disorders) | 1
TRANSIENT SQUEAK (General disorders) | 1
HAD TREE FALL ON BACK AND SHOULDER (General disorders) | 1
LUCENT FRACTURE (Musculoskeletal and connective tissue disorders) | 1
WORSENING OF RIGHT MCP AND CMCJ OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
"SQUEAKING" SOUND FROM JOINT OF RIGHT SHOULDER WITH MOVEMENT (Musculoskeletal and connective tissue disorders) | 1
PINS-AND-NEEDLES IN R THUMB/INDEX/MIDDLE FINGER, RADIATING TO ELBOW AND INTO R BREAST (Musculoskeletal and connective tissue disorders) | 1
VAGAL EPISODE (DIZZY / FAINTING) POST SURGERY SECONDARY TO PAIN (General disorders) | 1
TENDONITIS OF LEFT SHOULDER- CLICKING/PAINFUL SENSATION WITH SHOULDER MOVEMENT (Musculoskeletal and connective tissue disorders) | 1
PAIN AND WEAKNESS IN RIGHT SHOULDER WHEN OVERWORKED. (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF TENDINOPATHY OF RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
SQUEAKING SOUND IN LEFT SHOULDER / PYROTITAN WITH MOVEMENT OF SHOULDER (Musculoskeletal and connective tissue disorders) | 1
PERSISTENT PAIN IN ANTERIOR LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
OCCASIONAL SQUEAK FROM IMPLANT. NOT PAINFUL (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF DYSFUNCTION IN RIGHT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
LEFT SIDED FORAMINA STENOSIS AT C5 AND C6 (Musculoskeletal and connective tissue disorders) | 1
INCREASED GRINDING/CLICKING IN LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
NERVE DISTURBANCE IN DISTRIBUTION OF MUSCULOCUTANEOUS NERVE AND/OR C6/C7 (Nervous system disorders) | 1
SQUEAK IN RIGHT SHOULDER JOINT WITH MOVEMENT (Musculoskeletal and connective tissue disorders) | 1
MINIMAL INFERIOR OSTEOPHYTE GLENOID. - XR + MRI REPORT. (Musculoskeletal and connective tissue disorders) | 1
ASYMPTOMATIC MARKED SUBARTICULAR CYSTIC CHANGES INVOLVING MID AND SUPERIOR GLENOID (Musculoskeletal and connective tissue disorders) | 1
SQUEAKING NOTED BY PATIENT FROM LEFT SHOULDER (Musculoskeletal and connective tissue disorders) | 1
SUBCORTICAL CYST IN POSTERIOR GLENOID INCREASED IN MEASUREMENT (UP TO 11MM) (Musculoskeletal and connective tissue disorders) | 1
DIFFICULTY IMPLANTING (DIFFICULTY BROACHING, REAMING AND INSERTING) (Musculoskeletal and connective tissue disorders) | 1
OCCASSIONAL SQUEAK NOTED IN OPERATIVE SHOULDER (Musculoskeletal and connective tissue disorders) | 1
FELL ONTO A OUTSTRETCHED ARM. NOW PAINFUL, TIGHT IN DELTOID REGION (Musculoskeletal and connective tissue disorders) | 1
PROSTHETIC LOOSENING (General disorders) | 1
FALL OFF BACK OF CAMPING BUS 1.5 METRES (Musculoskeletal and connective tissue disorders) | 1
RADIAL NERVE PALSY (Nervous system disorders) | 1
ANTERIOR DELTOID ATROPHY MODERATE STIFFNESS (Musculoskeletal and connective tissue disorders) | 1
NERVE PAIN AND MILD LOSS OF SENSIBILITY IN DIGITS 1 AND 2 LEFT HAND (Nervous system disorders) | 1
SUFFERED A FISSURE FRACTURE COLLUM CHIRURGICUM LEFT SIDE. (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was managed by Ascension Orthopedics, Inc prior to Smith+Nephew Inc. (Memphis) becoming the sponsor in January 2021. This study was not designed nor controlled/monitored by Smith+Nephew Inc. (Memphis), except for the final follow-up phase. The data reported is based on the data available since the time of Smith+Nephew's acquisition of Ascension Orthopedics, Inc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period up to 60 days but less than or equal to 120 days from the time submitted to the sponsor for review. Sponsor may delay publication up to 120 days to permit the filing of appropriate patent applications if the sponsor believes any publication contains any information relating to patentable items and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2013-05-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT02405208/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT02405208/SAP_001.pdf